CLINICAL TRIAL: NCT00936533
Title: Botulinumtoxin A Treatment in Epidermolysis Bullosa Simplex and Pachyonychia Congenita - a Double-blind Placebo-controlled Phase II Proof of Concept Study
Brief Title: Botulinumtoxin A Treatment in Epidermolysis Bullosa Simplex and Pachyonychia Congenita
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Dr Carl Swartling, Sophiahemmet
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBSBTXA09; EudraCT number 2009-010763-17
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Epidermolysis Bullosa Simplex
MeSH Terms: conditions — Epidermolysis Bullosa Simplex | interventions — abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dysport® (Botulinumtoxin A (Btx A)) — Single injection in patients´ soles with Btx A in one foot and sodium chloride in the other, with the possibility of a second injection after 12 weeks. The drug will be given in general anaesthesia after curettage of the focal hyperkeratoses. Only the areas with focal hyperkeratoses will be injected with 50 ul per injection.The active drug Btx A (Dysport®, solution for injection) has a concentration of 100 U/ml, and the maximum dose is 300 U per foot.
  Other Names: Dysport®
Drug: Placebo — Placebo preparation without active compound, administered as the active drug.
  Other Names: Dysport Placebo

SUMMARY:
This study evaluates the clinical effect of foot injection of the bacteria protein Botulinum toxin A on plantar pain in patients with EBS (epidermolysis bullosa simplex) or PC (pachyonychia congenita).

DETAILED DESCRIPTION:
Epidermolysis bullosa simplex (EBS) is the most common subtype of epidermolysis bullosa and mutations in keratin genes (KRT 5/14) are responsible for this condition. Painful blisters and keratoderma of the feet are common and the blisters in EBS typically get worse in the summer due to sweating and increased environmental heat. Since 2010, also the related condition pachyonychia congenita (PC) is included in the study. The primary objective of the study is to evaluate the clinical effect of Botulinum toxin A (Dysport®), injected in the foot, on plantar pain in patients with EBS or PC. Quality of life, pain in feet, effect duration, plantar sweating and safety of the treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent received from patient
* Informed consent received from patient´s parents (when patient < 18 years)
* A solid EBS-diagnosis based on genetic analysis and/or phenotype. The EBS-diagnosis will be performed by Professor Anders Vahlquist, Swedish Centre of Genetic skin disorders, Uppsala.
* Age > 16 years
* Patients must be previously untreated with Btx A
* If female, patient is post-menopausal, surgically sterilized, or willing to use an acceptable method of birth control

Exclusion Criteria:

* Contraindication to Btx A
* Contraindication to general anaesthesia
* Use of aminoglycosides, tetracyclines , spectinomycin, lincomycin, polymyxin or muscle relaxants
* Pregnancy or lactation
* Patients unwilling to meet the requirements of the protocol
* Other medical or social reasons for exclusion at the discretion of the Investigator

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Determination of the difference between treated and untreated foot in change of pressure (measured by manometry) to reach unbearable pain, VAS=8, from baseline to 5 week after injection. | 5 weeks

SECONDARY OUTCOMES:
Quality of life using a questionnaire (DLQI) | 12 or 17 weeks
Pain in feet using a questionnaire (VAS) | 5, 12 (and 17) weeks
Effect duration measured with manometry (same as primary end-point but measured at week 12) | 12 weeks
Safety by recording of reported adverse events (AE) by the patient at the clinic visits | 5, 12 (and 17) weeks
Foot-sweating using iodine-starch imprints before and after injections | 0 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carl Swartling, Principal Investigator — Uppsala University
Locations (1):
- Svettmottagningen, Sofiahemmet, Stockholm, Sweden